CLINICAL TRIAL: NCT01251497
Title: ¡Si, Yo Puedo Control Mi Diabetes!: A Diabetes Self-management Education Program for Hispanic/Latinos
Acronym: Yo Puedo
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas AgriLife Extension Service (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Ninfa Pena-Purcell, PhD, CHES, Texas AgriLife Extension Service, Texas A&M University System
Model: Parallel | Purpose: Supportive Care
Other Study IDs: texn0043
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes, Hispanic/Latinos, Diabetes Self-management Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: diabetes self-management education

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the íSi, Yo Puedo Controlar Mi Diabetes! (Yo Puedo) diabetes self-management education program.

ELIGIBILITY:
Inclusion Criteria: Self-identification as Hispanic/Latino, over the age of 18 years of age, diagnosis of type 2 diabetes and willingness to participate in the diabetes self-management education class.

Exclusion Criteria: non-diabetic persons, non English-speaking Hispanic/Latinos with type 2 diabetes

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)